CLINICAL TRIAL: NCT03857698
Title: The Effect of Body Stabilization Exercises on Balance, Functional Performance and Lumbar Lordosis Angle in Patients With Total Knee Prosthesis: Randomized Controlled Double Blind Study
Brief Title: The Effect of Body Stabilization Exercises on Balance, Functional Performance and Lumbar Lordosis Angle in Patients With Total Knee Prosthesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20190105
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: Total Knee Prosthesis; Stabilization Exercise; Balance; Functional Performance; Lumbar Lordosis Angle

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Evaluation of pain (Experimental): The patient's pain will be evaluated by VAS (visual analog scale) at the end of the treatment, at the end of the treatment and at the end of the 3 months follow-up. For this, a 10 cm long line will be drawn. 0: painless and 10: the most severe pain is described and the patient will be asked to mark the value corresponding to the pain (rest, activity and night pain) on the scale.
  Interventions: Other: Conservative Physical Therapy; Other: Body Stabilization Exercise
- Evaluation of joint range of motion (Experimental): The flexion and extension range of motion of the knee joints of the patient will be measured in the prone position using a universal goniometer before and after the training.
  Interventions: Other: Conservative Physical Therapy; Other: Body Stabilization Exercise
- Assessment of balance (Experimental): Postural stability will be evaluated by a Prokin brand balance device (ProKin, Tecnobody, Bergamo, Italy), a force platform. After the tests are explained to the patients, the physical characteristics of the patients (age, height, body weight) will be recorded on the device and the device will be calibrated. The patients' feet will be placed naked on the platform with reference to the lines on the x and y axis. During the test, the arms will be in free position near the body. The tests will be performed on both feet with both eyes open and eyes closed. Each test will last 30 seconds. After each test has been completed, the device will be recalibrated. As a result of the tests, the ellipse area (mm2) and perimeter (mm) parameters will be recorded for statistical analysis. In addition, the patient's stability limits will be calculated as a percentage.
  Interventions: Other: Conservative Physical Therapy; Other: Body Stabilization Exercise
- Evaluation of functional performance (Experimental): A timed up and go test is a test that assesses the mobility and lower extremity mobility. For this test, the patient will be asked to lift from a chair with armrest (sitting height: 46 cm), walk 3 meters as fast as possible, turn around the colored band marked on the floor and sit in the same chair. The elapsed time for the motion will be recorded in seconds.
  Interventions: Other: Conservative Physical Therapy; Other: Body Stabilization Exercise
- Lumbar lordosis angle assessment (Experimental): During the test, patients will be asked to stand upright in a comfortable position. In the evaluation of the lumbar lordosis, the inclinometer will first be fixed to the T12-L1 backbone and then to the L5-Sl backbone and the angular values in both measurements will be collected and recorded as lordosis angle.
  Interventions: Other: Conservative Physical Therapy; Other: Body Stabilization Exercise
- Evaluation of knee functionality (Experimental): It will be measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). There are three subgroups, namely pain, stiffness and function. A total of 24 questions (pain 5 questions, 2 questions of malfunction and 17 questions of function) and the scale answered by patients are completed in approximately 5 minutes. The scale is a 5-point Likert-type scale (0 = none 1 = mild 2 = moderate 3 = severe 4 = very severe). The score range for the subgroup of pain is 0-20, for the subgroup group 0-8 and for the subgroup of function is 0 - 68. The total WOMAC score is obtained by the sum of these 3 points and the maximum total WOMAC score is 96. There is a linear ratio between the scores obtained from the WOMAC index and the presence of symptoms. The high scores were associated with severe symptoms, more disability and poor health status, whereas low scores indicated that symptoms, pain, and functionality were good.
  Interventions: Other: Conservative Physical Therapy; Other: Body Stabilization Exercise
- Assessment of lower extremity muscle endurance (Experimental): The patient will be asked to sit on the chair as fast as possible, so that the chair, which has a 46 cm height, will be crossed in the chest. The stopwatch is started with the command given to the patient and stopped in 30 seconds. The number of repetitions will be recorded.
  Interventions: Other: Conservative Physical Therapy; Other: Body Stabilization Exercise

INTERVENTIONS:
Other: Conservative Physical Therapy — Patients who were discharged from the hospital and received the sutures will be supervised 2 days a week for 8 weeks. Exercise programs will be promoted individually.
  * Ice application for pain, edema control
  * Patellar mobilization
  * Three-way straight leg lifting exercises
  * Isometric exercises around the hips and knees
  * Active assisted, active, resistant knee range of motion exercises
  * Heel shift exercises in supine and sitting
  * Hip abduction on the side lying
  * Stretching exercises for patients with gastrosoleus, hamstring, hip flexor muscles
  * Neuromuscular Electrical Stimulation (NMES) for quadriceps muscle of patients will be applied. The isometric quadriceps contraction observed during the procedure will be required to actively participate in the patients.
Other: Body Stabilization Exercise — In the first session, breathing control and alet abdominal hallawing of movement will be taught to the patients with the help of the pressure biofeedback device. The degree of difficulty of the exercises will be improved by using different positions, by adding rotations to the motion, making the pelvic control more difficult and increasing the number of repetitions. In case of exacerbation of symptoms, the level will not be advanced. Exercises will be advanced according to the patient's initial level and response to exercise.
  * Consecutive shoulder flexion and extension in supine
  * Building a bridge
  * Lower body and hip flip
  * Single leg extension with bilateral arm elevation
  * Resilient leg stretch with bilateral arm elevation
  * Hip external rotation in lateral hospitalization
  * Side-lying arm opening
  * Shoulder girdle retraction on ball, horizantal abduction and extension

SUMMARY:
The aim of the study was to compare the efficacy of body stabilization exercises to be applied in addition to conservative physical therapy in patients undergoing total knee arthroplasty. Through this study, we aim to contribute to the literature and the clinic with objective, evidence-based results.

Ostetoarthritis includes the entire joint in a disease process involving the loss of articular cartilage in focal and progressive hyaline, including the increase in osteophytes and the thickness of the subchondral bone. Clinical symptoms of osteoarthritis include joint stiffness, pain, and dysfunction. Knee osteoarthritis causes activity limitation especially in the elderly. American Society of Orthopedic Surgeons, nonsteroidal anti-inflammatory drugs or tramadol in the medical treatment of osteoarthritis; they recommend reinforcement in conservative treatment, low intensity aerobic exercises and neuromuscular training programs. Total knee arthroplasty is preferred for surgical treatment to reduce pain, improve deformity, and improve functional range and range of motion in patients with advanced stage osteoarthritis who do not respond to conservative treatment. Total knee arthroplasty is a surgical procedure in which an artificial joint replaces the damaged knee joint. After knee arthroplasty, there was a decrease in pain, increased range of motion and improved quality of life.

Patients with osteoarthritis have a decrease in proprioceptive sensation due to inflammation in the knee joints and a decrease in knee mechanoreceptors. In addition to this proprioceptive disorder, muscle weakness caused by aging, decreased vision and losses in the central nervous system cause balance effects. This effect of equilibrium increases the fear of falling in individuals and therefore patients tend to move less. Therefore, the resulting inactivity causes a decrease in endurance with muscular force and causes the patients to become more immobile. This is particularly a risk factor for falls in patients with symptomatic lower extremity osteoarthritis and these causes mortality and morbidity.

Lumbopelvic-hip complex or "core" in lumbar vertebrae, pelvis, hip joints and active and passive structures that produce or restrict the movement of these segments. Core stability is associated with lower extremity balance performance. Body stabilization exercises decrease the risk of falling patients and improve their balance. Although stabilization exercises are performed in patients with total prosthesis in the literature, there is no study evaluating the effectiveness of these exercises on balance, functional performance and lumbal lordosis angle.

DETAILED DESCRIPTION:
A prospective, randomized controlled, double-blind clinical study was performed in unilateral total knee arthroplasty (TDP) surgery with a cross-linking, fixed insert, cemented total knee prosthesis and the same type of surgical technique. Ankara Yenimahalle Training and Research Hospital Patients admitted to the Rehabilitation Policlinic will be included in the study. Pre-study volunteers will be randomly assigned into two groups by giving information about the purpose and content of the study. The participants will be evaluated by a blind researcher before, after and 3 months after the treatment and the data obtained from the evaluation results will be analyzed by appropriate statistical methods.

Patients who have at least 80 degrees of knee flexion and full knee extension, who can be mobilized (with ancillary equipment), who can go up and down the stairs, without any infections, will be included in the study after their sutures have been taken. Patients will be randomly divided into two groups as education group and control group. The patients in the control group will undergo a conservative physical therapy program under the supervision of the physiotherapist. The patients in the training group will be given conservative treatment and body stabilization exercise program under the supervision of physiotherapist. The assessments before and after the treatment and after 3 months will be performed by another physiotherapist who does not know what treatment the patients are receiving. Pre-treatment, post-treatment and 3-month post-treatment pain with visual analog scale, joint motion range with goniometer, functional performance with time up and go test, balance with Prokin balance device (ProKin, Tecnobody, Bergamo, Italy), lumbal lordosis angle with Baseline Bubble Inclinometer®, knee functions with Western Ontario and McMaster Universities Osteoarthritis Index, the lower extremity muscle endurance with 30 second chair stand test will be evaluated. Patients in both groups will be treated for a total of 8 weeks 2 days a week.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Unilateral Total Knee Prosthesis Patients with full knee extension Patients with at least 80 degrees of knee flexion Mobilized (with ancillary equipment) Patients who can climb up and down stairs Patients who are not at risk for cardiac performance in terms of exercise and evaluation tests

Exclusion Criteria:

* Another musculoskeletal problem that may affect lower limb performance A neurological or oncological disease that affects the balance Limb length difference of more than 5 cm before or after surgery Patients with any systemic problem Patients with infection in the knee after surgery

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of functional performance | 10 months
  A timed up and go test is a test that assesses the mobility and lower extremity mobility.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Esenboğa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No